CLINICAL TRIAL: NCT06661525
Title: Advanced Optical Monitoring of Free Tissue Transfer Hemodynamics
Brief Title: Monitoring Free Tissue Transfer Hemodynamics Using NIRS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Surrey Memorial Hospital (SMH) (Unknown); Vancouver General Hospital (Other)
Responsible Party: Principal Investigator, Donald W. Anderson, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H22-03706
Record Dates: First submitted 2024-05-02; First posted 2024-10-28 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Oxygen Supply Absent
Keywords: NIRS Sensor; Tissue Oxygenation; Free Tissue Transfer (FTT)
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Participants (Experimental): Data collection from Participants and evaluate their feedback by filling a questioner
  Interventions: Device: Free Flap NIRS
- Care providers (Active Comparator): Care providers will provide their feedback via questioner
  Interventions: Device: Free Flap NIRS

INTERVENTIONS:
Device: Free Flap NIRS — Monitoring of tissue oxygenation after Free Tissue Transfer (FTT) surgeries.

SUMMARY:
Free tissue transfer (FTT) is a surgical procedure for repairing cancer resection wounds. Free tissue transfer usually involves taking skin from one area of the body (e.g. leg) and transplanting it to the surgically created wound (e.g. neck wound). Due to problems with anastomosis, the transplanted skin can die. If the poor blood supply can be detected early, transplanted skin can be saved by taking patients back to the operating room. The investigators propose to improve the design and test a novel, non-invasive monitoring system specifically for head and neck surgeries for early detection of poor blood supply to the transplanted tissue after FTT surgery.

DETAILED DESCRIPTION:
PURPOSE: To improve the design and evaluation of a novel spatially resolved near-infrared spectroscopy (NIRS) system customized for continuous postoperative free tissue transfer (FTT) monitoring and to make this system commercially available.

HYPOTHESIS: The novel NIRS device is capable of monitoring FTT reconstruction continuously for 72 hours after surgery with minimal interference to patient care, minimal discomfort to the patient, and minimal interference with clinical assessment.

JUSTIFICATION FOR THE STUDY: FTT consists of transplanting skin, muscle or bone along with its feeding blood vessels from one body site to reconstruct a defect created by removing cancerous tumours or traumatic injury at a separate site. The key to the survival of the transplanted tissue is the meticulously created microvascular anastomosis between the blood vessels of the transplanted tissue and the blood vessels of the recipient site. Microsurgical techniques have been refined over time to maintain the patency of the anastomosed blood vessels. Nevertheless, the current FTT failure rate is between 1 and 10%.

When FTT failure occurs, it is a devastating experience for the patient and the surgical team. The patient has to be urgently brought to the operating room for an attempted salvage of the microvascular anastomosis. In the event of unsuccessful salvage, the patient has to undergo multiple surgeries that compound the associated morbidity, prolong hospital stay, and increase health care costs. Early detection of vascular compromise is essential for increasing the odds of successful salvage. Thus, the methods used to monitor the FTT vascular status are critical and have received much attention in the literature. Clinical examination remains the gold standard and the most popular method of monitoring FTT viability. The two downsides of clinical examinations are the requirement for personnel trained and experienced in FTT monitoring and the inability to provide reliable continuous monitoring. Therefore recognition of FTT compromise is often delayed significantly compromising successful surgical salvage attempts.

Recently, NIRS has been recognized as the technology with the most potential to address the problems seen with FTT clinical monitoring. NIRS is a non-invasive technique that passes near-infrared light (600-1000 nm) through the tissues at a depth of 10 to 20 mm. Calculating the amount of absorbed light allows real-time measurements of oxygenated, deoxygenated, and total hemoglobin concentrations. Therefore, an abnormality of tissue perfusion and oxygenation can then be detected instantaneously and confirmed clinically. Reducing the time from detection of vascular compromise to the attempted FTT rescue in the operating room decreases the ischemia time and increases the FTT salvage rate.

A recent meta-analysis concluded that NIRS is "a reliable monitoring technique that is non-invasive, objective, and easy to use". However, there are currently no NIRS systems available that can monitor FTT used in head and neck surgery. This is largely due to the difficulty in creating NIRS sensors that are small enough to be used in the head and neck region. Developing and evaluating a novel, customized NIRS system with a miniaturized sensor suitable for a variety of FTT options is needed, presenting an attractive clinical opportunity.

The proposed study's principal investigator (D.W.A.) is the pioneer of head and neck FTT in British Columbia, with FTT experience spanning over 35 years. He will use his expertise to consult with Dr. Shadgan, a clinical biophotonics research scientist, to provide clinical and technical specifications required for the construction of the NIRS prototype. Currently, they successfully built and tested the miniaturized NIRS sensor on 3 patients, and they were able to obtain promising results. To establish our method and refine the design of the sensor to be compatible with a wide variety of FTT surgeries, The investigators plan to conduct this pilot study.

OBJECTIVES

1. Develop a novel NIRS system with miniaturized sensors suitable for various FTT reconstruction options.
2. Conduct a pilot study on up to 60 patients to determine perfusion thresholds indicative of vascular compromise for a variety of FTT reconstructive options, and to improve the design and application of sensors to the variety of FTT.

RESEARCH DESIGN

The NIRS prototype will be tested intra- and post-operatively on a single patient undergoing FTT reconstruction. Intra-operative NIRS measurements simulating FTT compromise will be collected during a single FTT operation.

Post-operatively the NIRS probe will be placed and fixed over the FTT for 72 hours and its measurements will be recorded. In addition, experienced nurses not involved in the proposed study will monitor the FTT vascular status with the conventional clinical methods currently employed at VGH and Surrey Memorial Hospital. The clinical assessment will be documented in the standardized table and correlated to the NIRS recordings. Finally, at the end of the 72-hours, both the patient and the clinicians will complete questionnaires to evaluate their experience with the NIRS system.

STATISTICAL ANALYSIS

The collected intra-operative and post-operative NIRS measurements will be used to establish a threshold for low perfusion alarm on the NIRS monitor for different types of tissues.

The data that will be collected through patients' and doctors' questionnaires will go through descriptive statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* 60 patients undergoing a variety of free tissue transfer for head and neck cancer. The result of the reconstruction should be easily visible to the clinicians.
* Age of 18 years old or older

Exclusion Criteria:

* Serious medical condition or other disease which occurs at the same time
* Metastatic disease
* Pregnant or nursing

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-20 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Establish a baseline Total Oxygenation Index (TOI) to measure NIRS on FTT cases | Up to 36 months
  The total oxygenation index (TOI) measurements will be used to establish a TOI baseline for Free Tissue Transfer (FTT) and to calibrate and tune the FTT-system
Enhance the design and accuracy of the FTT- NIRS sensor based on patient and clinicians feedback | 24 months
  The data collected will be used to enhance the design and accuracy of the next generation of NIRS sensors based on the feedback provided by the patient and clinician

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Surrey Memorial Hospital, Surrey, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No